CLINICAL TRIAL: NCT01352351
Title: Linking Microcredit, Technology, and Promotion of IYCF Breastfeeding Guidelines in Bauchi State, Nigeria
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: University of California, Davis (Other); Partners for Development (Unknown); The Alive & Thrive Small Grants (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 11-0534
Record Dates: First submitted 2011-05-10; First posted 2011-05-11 (Estimated); Last update posted 2013-02-08 (Estimated); Status verified 2013-02

CONDITIONS: Breast Feeding Exclusive; Initiation of Breastfeeding
Keywords: Breast feeding Exclusive; Initiation of breastfeeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Breastfeeding promotion intervention (Experimental): Intervention:
  * Group breastfeeding counseling during monthly microcredit borrower group meetings
  * Weekly cell phone messages about breastfeeding
  Interventions: Behavioral: Breastfeeding promotion intervention
- No intervention (No Intervention): The no intervention group will participate in their regular microcredit borrower group meetings, but will not receive breastfeeding counseling or cell phone messages.

INTERVENTIONS:
Behavioral: Breastfeeding promotion intervention — * Breastfeeding counseling during monthly microcredit meetings
  * Weekly cell phone messages about breastfeeding
  Arms: Breastfeeding promotion intervention

SUMMARY:
The University of North Carolina (UNC) and Partners for Development (PFD), an American non-governmental organization, will conduct a 2-year cluster-randomized controlled trial in Bauchi State, Nigeria, to test the effectiveness of two behavior change strategies for increasing the proportion of participants who exclusively breastfeed their infants until 6 months. The investigators will build upon PFD's existing microcredit and reproductive health program by adding face-to-face breastfeeding education during borrowers' meetings and bi-weekly cell phone breastfeeding messages. The hypothesis is that the control group will remain at the baseline level for exclusive breastfeeding to 6 months, while the intervention group will increase by 15%. The investigators will measure the effectiveness of the intervention by conducting baseline and final surveys with a cohort of 485 female borrowers who are pregnant at time 1 and who have a 6-month-old infant at time 2. The data will be analyzed using logistic regression adjusting for possible confounders and the effect of clustering.

ELIGIBILITY:
Inclusion Criteria:

* Participation in a microcredit borrower group sponsored by Partners for Development in Bauchi, Dass, or Ganjuwa Local Government Authority in Bauchi State, Nigeria
* Female (15-45 years)
* Pregnant at baseline

Exclusion Criteria:

* Female (<15 years)
* Not pregnant

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 485 (Actual)
Dates: Start 2011-05; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Proportion of women who exclusively breastfeed to 6 months | The outcome will be measured when the infant is 6-7 months old.

SECONDARY OUTCOMES:
Proportion of women who exclusively breastfeed for 0-1 month | The outcome will be measured when the infant is 6-7 months old.
Proportion of women who exclusively breastfeed for 2-3 months | The outcome will be measured when the infant is 6-7 months old.
Initiation of breastfeeding within 1 hour of birth | The outcome will be measured when the infant is 6-7 months old.
Proportion of infants who receive pre-lacteal feeds | The outcome will be measured when the infant is 6-7 months old.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret E. Bentley, PhD, Principal Investigator — Carolina Population Center, University of North Carolina at Chapel Hill; Valerie L. Flax, PhD, Principal Investigator — Carolina Population Center, University of North Carolina at Chapel Hill; Mekebeb Negerie, DrPH, Principal Investigator — Partners for Development/Nigeria

REFERENCES:
- [Derived] Flax VL, Negerie M, Ibrahim AU, Leatherman S, Daza EJ, Bentley ME. Integrating group counseling, cell phone messaging, and participant-generated songs and dramas into a microcredit program increases Nigerian women's adherence to international breastfeeding recommendations. J Nutr. 2014 Jul;144(7):1120-4. doi: 10.3945/jn.113.190124. Epub 2014 May 8. PMID 24812071